CLINICAL TRIAL: NCT01370954
Title: NAC-003 P.L.U.S. Program (Progress Through Learning Understanding & Support)
Status: Completed | Type: Observational
Sponsor: Pamlab, Inc. (Industry)
Collaborators: InfoMedics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NAC-003
Record Dates: First submitted 2011-05-20; First posted 2011-06-10 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Early Memory Loss; Mild Cognitive Impairment; Alzheimer's Disease; Vascular Dementia
Keywords: CerefolinNAC; early memory loss; pre-alzheimer's disease; cognitive function; folic acid; folate; L-methylfolate; vitamin B12; methylcobalamin; N-acetylcysteine; NAC; oxidative stress; memory deficit; antioxidant
MeSH Terms: conditions — Memory Disorders; Cognitive Dysfunction; Alzheimer Disease; Dementia, Vascular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CerefolinNAC®: Subjects diagnosed with Early Memory Loss who have been prescribed CerefolinNAC® daily.
  Interventions: Other: CerefolinNAC®

INTERVENTIONS:
Other: CerefolinNAC® — CerefolinNAC® is an orally-administered medical food, and each caplet contains 2 mg Methylcobalamin, 600 mg N-acetylcysteine, and 6 mg of L-methylfolate Calcium (as Metafolin®), which is the primary biologically active and immediately bioavailable form of folate. Dosage will be 1 caplet QD.

SUMMARY:
This study will be an observational study in which patients who have been prescribed CerefolinNAC® are invited to participate in surveys regarding their experiences with CerefolinNAC®. CerefolinNAC® is a medical food indicated for the distinct nutritional requirements of individuals under treatment for early memory loss with particular emphasis for those individuals diagnosed with or at risk for neurovascular oxidative stress and/or hyperhomocysteinemia; mild to moderate cognitive impairment with or without vitamin B12 deficiency, vascular dementia or Alzheimer's disease. The purpose of this study is to increase the understanding of the role of CerefolinNAC® in managing proper neuronal function in the brain, provide patients with personalized education and support, and contribute to the overall understanding of the needs and concerns of patients being treated for early memory loss.

DETAILED DESCRIPTION:
Surveys used to conduct this study will be administered via telephone by InfoMedics, Inc., a company with an established system for developing such patient-physician feedback programs. Participating physicians will ask their patients to participate in the program after CerefolinNAC® has been prescribed and provide them with a brochure containing an introduction to the program and instructions on how to enroll. Patients self-enroll, take a brief survey before starting their CerefolinNAC® prescription, and then two brief follow-up surveys at 6 weeks and 12 weeks. As patients complete surveys within the study, their physician will receive individualized feedback reports outlining their patient's treatment experience and progress. Patients will also receive a copy of their own reports, to help encourage them to continue taking CerefolinNAC® as directed. Patients will also receive educational materials about managing their early memory loss.

ELIGIBILITY:
Inclusion Criteria:

* New CerefolinNAC® Start
* Only for patients who have been prescribed CerefolinNAC® to help metabolic management of early memory loss.

Exclusion Criteria:

* If a participant indicates that he or she did not get a prescription for CerefolinNAC®, he/she will not be able to complete the survey(s).
* For follow-up surveys, if the participant indicates that he/she has not been taking CerefolinNAC®, he/she will not be able to complete the survey (s).

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Early Memory Loss Who Have Been Prescribed CerefolinNAC®
Sampling Method: Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To determine if CerefolinNAC® affects a subject's quality of life as measured by the Quality of Life-Alzheimer's Disease Scale (QOL-AD) | Baseline, Week 6 and Week 12
  The QOL-AD is a brief, 13-item measure designed specifically to obtain a rating of the patient's Quality of Life.

SECONDARY OUTCOMES:
To determine overall patient satisfaction with CerefolinNAC® using a 9-point satisfaction scale | Weeks 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Donald E Schmechel, M.D., Principal Investigator — Falls Neurology and Memory Center
Locations (1):
- Falls Neurology and Memory Center, Hickory, North Carolina, United States